CLINICAL TRIAL: NCT00795990
Title: Timing for the Medical Treatment of Patent Ductus Arteriosus in Preterm Infants
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Carrie Rau, University of Utah
Other Study IDs: 31769
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Patent Ductus Arteriosus
Keywords: Efficacy of early vs late use of ibuprofen for PDA closure
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective chart review to look at the timing of using indomethacin and ibuprofen for PDA closure for infants admitted into the NICU of the University of Utah Hospital from 1/2007-8/2008. The purpose is to compare the outcomes of medical intervention in preterm infants if intervention occurs day of life 4 or less, or day of life 5 or greater, with the birthdate being counted as day of life 1.

DETAILED DESCRIPTION:
This is a retrospective chart review to look at the timing of using indomethacin and ibuprofen for PDA closure for infants admitted into the NICU of the University of Utah Hospital from 1/2007-8/2008. The purpose is to compare the outcomes of medical intervention in preterm infants if intervention occurs day of life 4 or less, or day of life 5 or greater, with the birthdate being counted as day of life 1. All infants born less than 1200 gms will be evaluated for whether or not an echocardiogram was done. If an echocardiogram was done that showed a PDA, data will be collected as to what medical interventions were done, at what age, and what were the results of the medical intervention. Infants will be stratified into birthweights <800 gm and 800-1200 gm.

ELIGIBILITY:
Inclusion Criteria:

* birth weight less than 1200 gm

Exclusion Criteria:

* none

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants born weighing less than 1200 gms with echo confirmed PDA
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2008-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Early versus Late Medical Treatment of PDA | 1 month
  The primary objective is to compare early (day of life 4 or less) versus late (day of life 5) medical treatment of PDA. Data will be collected via a retrospective chart review. Information will be collected on both the use of indomethacin and ibuprofen. Both medications are used as standard of care in the NICU for closure of PDAs.

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Chan, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States